CLINICAL TRIAL: NCT02350790
Title: Robotic Surgical Management of Endometriosis: Excision Versus Ablation With Argon Beam Coagulator (ABC)
Brief Title: Robotic Surgical Management of Endometriosis: Excision Versus Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Timothy A Deimling, Assistant Professor, Division of Obstetrics and Gynecology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 43830
Record Dates: First submitted 2013-08-20; First posted 2015-01-30 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Endometriosis
Keywords: Robotics; Laparoscopy; Endometriosis; Argon; Gynecology
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic ablation (Active Comparator): Half of the patients in the study will be randomized to robotic ablation of endometriosis with the argon beam coagulator (ABC).
  Interventions: Procedure: Robotic ablation
- Robotic Excision (Active Comparator): Half of the patients in the study will be randomized to robotic excision of endometriosis.
  Interventions: Procedure: Robotic excision

INTERVENTIONS:
Procedure: Robotic ablation — Robotic laparoscopic ablation of endometriosis with the argon beam coagulator (ABC)
  Arms: Robotic ablation
Procedure: Robotic excision — Robotic excision of endometriosis
  Arms: Robotic Excision

SUMMARY:
Patients who are planning to undergo laparoscopic surgery for endometriosis will be assigned to either ablation or excision of endometriosis. The investigators think that patients who have excision of endometriosis will have greater relief of pain.

DETAILED DESCRIPTION:
Patients with known endometriosis based on prior surgical pathology or suspected endometriosis based on symptomatology who plan on undergoing diagnostic laparoscopy will be offered enrollment in the study. They will complete preoperative pain assessments with the tools outlined above. At the time of diagnostic laparoscopy, patients found to have endometriosis will be staged according to the American Society of Reproductive Medicine guidelines. Patients with Stage 4 or deeply infiltrating endometriosis will be excluded from the study. At that point, the patients will be randomized in the operating room to either laparoscopic excision of endometriosis or laparoscopic ablation with the argon beam coagulator. Patients will be stratified according to the presence or absence of the Levonorgestrel-Intrauterine Device.

Pain assessments will be performed immediately postoperatively in the recovery area. Pain assessments will again be performed at 4 weeks, 6 months and 12 months. We will use the VAS pain scale and validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Endometriosis
* Chronic Pelvic Pain
* Stage 1-3 Endometriosis
* Reproductive aged women

Exclusion Criteria:

* Stage 4 Endometriosis
* Deeply Infiltrating Endometriosis
* Patients who decline surgical management of endometriosis

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline pre-operatively
  Patients will document their pain on a VAS.
Visual Analog Scale (VAS) | 6 months
  Patients will document their pain on a VAS.
Visual Analog Scale (VAS) | 12 months
  Patients will document their pain on a VAS.

SECONDARY OUTCOMES:
Quality of Life and Pain Questionnaires | 4 weeks,
  Patients will complete quality of life and pain questionnaires to document their responses to treatment.
Quality of Life and Pain Questionnaires | 6 months
  Patients will complete quality of life and pain questionnaires to document their responses to treatment.
Quality of Life and Pain Questionnaires | 12 months
  Patients will complete quality of life and pain questionnaires to document their responses to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin A Riley, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Hart R, Hickey M, Maouris P, Buckett W, Garry R. Excisional surgery versus ablative surgery for ovarian endometriomata: a Cochrane Review. Hum Reprod. 2005 Nov;20(11):3000-7. doi: 10.1093/humrep/dei207. PMID 16246860
- [Background] Daniell JF, McTavish G, Kurtz BR, Tallab F. Laparoscopic Use of Argon Beam Coagulator in the Management of Endometriosis. J Am Assoc Gynecol Laparosc. 1994 Aug;1(4, Part 2):S9. doi: 10.1016/s1074-3804(05)80894-1. PMID 9073672
- [Background] Wright J, Lotfallah H, Jones K, Lovell D. A randomized trial of excision versus ablation for mild endometriosis. Fertil Steril. 2005 Jun;83(6):1830-6. doi: 10.1016/j.fertnstert.2004.11.066. PMID 15950657
- [Background] Abbott J, Hawe J, Hunter D, Holmes M, Finn P, Garry R. Laparoscopic excision of endometriosis: a randomized, placebo-controlled trial. Fertil Steril. 2004 Oct;82(4):878-84. doi: 10.1016/j.fertnstert.2004.03.046. PMID 15482763
- [Background] Abbott JA, Hawe J, Clayton RD, Garry R. The effects and effectiveness of laparoscopic excision of endometriosis: a prospective study with 2-5 year follow-up. Hum Reprod. 2003 Sep;18(9):1922-7. doi: 10.1093/humrep/deg275. PMID 12923150
- [Background] Falcone T, Lebovic DI. Clinical management of endometriosis. Obstet Gynecol. 2011 Sep;118(3):691-705. doi: 10.1097/AOG.0b013e31822adfd1. PMID 21860303